CLINICAL TRIAL: NCT03777709
Title: The FAITH! Trial: A mHealth Intervention to Improve Cardiovascular Health Among African-Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-006846; 5R21MD013490 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2018-12-17 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Diseases; Physical Activity; Diet Modification; Lifestyle Factors
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The FAITH! App intervention includes a 10-week core series of multimedia education modules with a LS7 focus and other features including interactive self-quizzes, self-monitoring (diet/physical activity), and social networking. Participants will follow a weekly schedule of each module concentrating on each LS7 component. Personalized messages will be delivered to each participant 3-4 times weekly over the intervention phase through the app dashboard, text message, or email. The sharing board will be moderated weekly to foster discussion on behavior change influences and participant successes/challenges to healthy lifestyle. Participants will maintain app access for the duration of the study.
  Interventions: Behavioral: FAITH! App
- Delayed Intervention/Control (No Intervention): The delayed intervention group will not receive additional materials while under the "control" time point (intervention group within intervention/maintenance phases).

INTERVENTIONS:
Behavioral: FAITH! App — Participants allocated to the intervention arm will complete a 10-week, individual-tailored intervention program utilizing the FAITH! App to promote the AHA LS7 through health education and to increase awareness and skill development while enhancing self-efficacy, self-regulation, and social support for healthy behavior change.
  Arms: Intervention

SUMMARY:
The purpose of this project is to apply a community-based participatory research (CBPR) approach to rigorously refine and test the feasibility and preliminary efficacy of an existing cardiovascular (CV) health and wellness digital application (app) prototype to improve CV health according to the American Heart Association Life's Simple 7 (LS7) framework among African-American (AA) adults within faith communities. The investigators hypothesize that the app-based intervention will be feasible and improve LS7 among AAs from baseline to 6-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. African American race/ethnicity
2. 18 years or older
3. Own a smart phone
4. Have basic Internet navigation skills
5. Have at least weekly Internet access (i.e. at home, church, or other public access)
6. Have an active email address
7. Intake of fruits/vegetables less than 5 servings a day
8. No engagement in regular physical activity
9. Able to engage in moderate physical activity

Exclusion criteria:

1. Unable to walk up 2 or more flights of stair or walk more than 1 city block without assistance or stopping
2. Pregnant (due to associated hormonal and weight changes)
3. Visual/hearing impairment or mental disability that would preclude independent app use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess C Brewer, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Given the community-based participatory process, it was decided as an academic-community team, that individual participant data will not be available to other researchers from this historically marginalized population.

REFERENCES:
- [Derived] Brewer LC, Jenkins S, Hayes SN, Kumbamu A, Jones C, Burke LE, Cooper LA, Patten CA. Community-Based, Cluster-Randomized Pilot Trial of a Cardiovascular Mobile Health Intervention: Preliminary Findings of the FAITH! Trial. Circulation. 2022 Jul 19;146(3):175-190. doi: 10.1161/CIRCULATIONAHA.122.059046. Epub 2022 Jul 18. PMID 35861762
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through various methods including phone calls, flyers, email, social media, and pastor referrals from February 2020 to October 2020. In-person and virtual kickoff events were held for study overview and open discussion forums, and the study principal investigator recorded a promotional video detailing study requirements and participant expectations. Interested individuals completed an electronic "Participant Interest/Eligibility Form," submitted to the study team.
Units Other Than Participants: site
Period: Overall Study
Arm/Group | Intervention | Delayed Intervention/Control
Started | 41; 8 site | 44; 8 site
Completed | 34; 8 site | 42; 8 site
Not Completed | 7; 0 site | 2; 0 site

BASELINE CHARACTERISTICS:
Units Other Than Participants: site
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Delayed Intervention/Control | Total
Number analyzed (Participants) | 34 | 42 | 76
Number analyzed (site) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.9) | 52.1 (11.4) | 54.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Identify as African-American: Yes | 34 | 42 | 76
  Identify as African-American: No | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Missing | 0 | 4 | 4
  Single | 9 | 11 | 20
  Divorced | 3 | 7 | 10
  Widowed | 0 | 1 | 1
  Married or committed relationship | 22 | 19 | 41
Education Level [Count of Participants; unit: Participants]
  Missing | 0 | 4 | 4
  High school graduate or less | 4 | 4 | 8
  Some college | 9 | 14 | 23
  Technical or Associate's degree | 7 | 6 | 13
  College graduate or higher | 14 | 14 | 28
Employment Status [Count of Participants; unit: Participants]
  Missing | 0 | 4 | 4
  Employed, at least Part-Time | 26 | 30 | 56
  Unemployed | 4 | 2 | 6
  Retired | 4 | 6 | 10
Household Income Category [Count of Participants; unit: Participants]
  <$35,000 | 8 | 6 | 14
  $35,000-$49,999 | 3 | 11 | 14
  $50,000-$74,999 | 12 | 9 | 21
  >=$75,000 | 7 | 8 | 15
  Not disclosed | 4 | 8 | 12
Healthcare Insurance [Count of Participants; unit: Participants]
  Missing | 0 | 4 | 4
  Yes | 30 | 34 | 64
  No/Don't Know | 4 | 4 | 8
Has healthcare professional, seen on regular basis [Count of Participants; unit: Participants]
  Yes | 26 | 33 | 59
  No | 8 | 9 | 17
Health conditions as communicated by a healthcare professional [Count of Participants; unit: Participants]
  Weight 20 pounds or more over ideal weight for your height and build: No | 12 | 10 | 22
  Weight 20 pounds or more over ideal weight for your height and build: Yes | 22 | 32 | 54
  Weight 20 pounds or more over ideal weight for your height and build: Missing | 0 | 0 | 0
  High blood pressure: No | 13 | 16 | 29
  High blood pressure: Yes | 21 | 26 | 47
  High blood pressure: Missing | 0 | 0 | 0
  Diabetes: No | 21 | 33 | 54
  Diabetes: Yes | 11 | 9 | 20
  Diabetes: Missing | 2 | 0 | 2
  High cholesterol: No | 19 | 25 | 44
  High cholesterol: Yes | 15 | 17 | 32
  High cholesterol: Missing | 0 | 0 | 0
Current cigarette smoker [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 1
  No | 33 | 40 | 73
  Yes | 1 | 1 | 2
Electronic health literacy score [Mean (Standard Deviation); unit: units on a scale] — Sum of 8 items: 8 (low) to 40 (high)
  units on a scale | 24.7 (6.9) | 28.2 (5.4) | 27.9 (6.0)
Mobile technology/Internet use skills [Mean (Standard Deviation); unit: units on a scale] — Mean of 3 items: 1 = low skill to 5 = high skill
  units on a scale | 3.9 (1.3) | 4.1 (1.0) | 4.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Life's Simple 7 Composite Score Change
Description: Change from baseline Life's Simple 7 Composite Score at 6 month post-intervention The Life's Simple 7 Composite Score is adapted from the American Heart Association standards based on health assessment data and is a composite of each component (average BP from 3 readings, fasting lipid panel and glucose, height, weight, self-reported cigarette smoking status, dietary quality, and physical activity patterns). Point values are assigned to each component: 2 points for ideal, 1 point for intermediate, 0 points for poor. The total sum allows for a continuous measure of cardiovascular health ranging from poor to ideal (0-14 points). The final score will be categorized as 0-6 (poor), 7-8 (intermediate), 9-14 (ideal).
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants able to attend and complete in person health assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 24 | 31
units on a scale | 1.88 (1.85) | 0.74 (1.69)
Statistical Analysis 1: Comparison: Intervention vs Delayed Intervention/Control; Effect size of 1-unit difference in mean LS7 score was based on meta-analysis indicating each unit increase in mean LS7 metrics equates to a 19% and 11% reduction in CVD and all-cause mortality, respectively. Power calculations to estimate sample size: church goal of 16 churches (8/arm), with mean 5 participants/church (40/arm) to provide 80% power to detect 1.45 difference in average LS7 score change between groups (.01 intracluster correlation, and .5 coefficient of variation of church sizes); Test type: Superiority; p < 0.0001, Regression, Linear — unadjusted p-value; Mean Difference (Final Values) = 1.45, Standard Deviation 2 — A recruitment aim of 40 participants per church (16 churches, 8 per arm, mean of 5 participants per church) provides 80% power to detect a difference of 1.45 in mean LS7 score change between groups (effect size 0.73)

2. Primary Outcome: Blood Pressure Change
Description: Change from baseline blood pressure at 6 month post-intervention. (average of 3 sitting readings of systolic and diastolic pressures)
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants able to attend and complete in-person health assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 24 | 31
mmHg
  Systolic BP | -3.09 (11.61) | -7.25 (13.14)
  Diastolic BP | -0.53 (8.27) | -2.5 (11.85)

3. Primary Outcome: Fasting Glucose (Fingerstick)
Description: Change from baseline to 6 months post-intervention fasting glucose
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who adhered to protocol for fasting glucose.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 9 | 11
mg/dL | 2.89 (18.44) | 6.73 (10.64)

4. Primary Outcome: Fasting Lipid Panel
Description: Change in fasting lipid panel from baseline to 6 months post-interventio
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants able to attend and complete in-person health assessment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 27 | 34
mg/dL | -10.96 (25.88) | -17.74 (25.93)

5. Primary Outcome: BMI
Description: Change from baseline BMI at 6 months post-intervention
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants able to attend and complete in person health assessment.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 27 | 34
kg/m^2 | -0.16 (1.30) | 0.14 (2.24)

6. Primary Outcome: Smoking Status Category
Description: Change in the categorical score (poor, intermediate, ideal) of the smoking status LS7 component from baseline to 6 months. Poor = Current Smoker, Intermediate = Former Smoker (<1 year), Ideal = Never or Former (>1 year).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 30 | 38
Participants
  Missing | 0 | 1
  Poor | 1 | 1
  Intermediate | 1 | 9
  Ideal | 28 | 27

7. Primary Outcome: Smoking Status Category
Description: as for outcome 6
Time Frame: 6 Months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 30 | 38
Participants
  Missing | 0 | 1
  Poor | 1 | 0
  Intermediate | 1 | 0
  Ideal | 28 | 37

8. Primary Outcome: Dietary Quality (According to American Heart Association Guidelines by the Validated, Culturally Appropriate, Delta Nutrition Intervention Food Frequency Questionnaire-FFQ)
Description: Dietary quality was measured using a checklist of foods and beverages, self-reported by participants at baseline and 6 months post-intervention. Responses range from never to 2 or more times per day (responses: never, < once/month, once/month, 2-3 times/month, 1 time/week, 2 times/week, 3-4 times/week, 5-6 times/week, 1 time/day, 2 or more times/day). Nutrient intake was estimated via a computer software, multiplying reported food frequency by nutrient content, following by comparison to AHA guidelines.
  Healthy diet score include 5 components:
  1. fruits and vegetables, ≥4.5 cups/d
  2. fish, 2 or more 3.5-oz servings/wk
  3. fiber-rich whole grains (≥1.1 g fiber/10 g carbohydrate), 3 or more 1-oz-equivalent servings/d
  4. sodium, ≤1500 mg/d
  5. sugar-sweetened beverages, ≤450 kcal/wk.
  Each component equals 1 point, resulting in scores from 0 to 5, which are categorized as Poor (0-1), Intermediate (2-3), or Ideal (4-5). Higher scores indicated better dietary quality.
Time Frame: Immediate post-intervention
Population: Number of participants analyzed reflects number of participants who completed the online questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 30 | 37
score on a scale | 1.9 (1.2) | 1.4 (1.2)

9. Primary Outcome: Dietary Quality (According to American Heart Association Guidelines by the Validated, Culturally Appropriate, Delta Nutrition Intervention Food Frequency Questionnaire-FFQ)
Description: as for outcome 8
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed the online questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 29 | 38
score on a scale | 0.79 (0.86) | -0.08 (1.19)

10. Primary Outcome: Physical Activity Patterns (Minutes/Week of Moderate and Vigorous Intensity Physical Activity, Measured by the International Physical Activity Questionnaire-IPAQ)
Description: Change from baseline in the total minutes per week that a participant engaged in moderate and vigorous intensity physical activity at immediate post-intervention.
Time Frame: Immediate post-intervention
Population: Differences in overall analyzed and specific rows are due to unanswered/missing survey data from participants.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 24 | 27
minutes/week
  Total minutes vigorous activity in the past week | 91.8 (192.1) | 98.5 (129.3)
  Total minutes moderate activity in the past week: number analyzed (Participants) | 24 | 23
  Total minutes moderate activity in the past week | 168.6 (238.5) | 80.7 (90)

11. Primary Outcome: Physical Activity Patterns (Minutes/Week of Moderate and Vigorous Intensity Physical Activity, Measured by the International Physical Activity Questionnaire-IPAQ)
Description: Change from baseline to 6 months post-intervention in the total minutes per week that a participant engaged in moderate and vigorous intensity physical activity.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed the online questionnaire.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 20 | 23
minutes/week | 219.70 (396.73) | 76.09 (286.67)

12. Primary Outcome: Intervention Feasibility Measures - Participant Engagement With Tracking
Description: Participant engagement with weekly diet/physical activity tracking measured by number of times participant engaged with the tracking feature at immediate post-intervention.
Time Frame: Immediate post-intervention
Population: Number of participants analyzed reflects number of participants who utilized tracking features.
  Outcome for Arm 2 (Control/Delayed Intervention group) is not shown as this group did not have access to the FAITH! App and as such could not have participated in the described outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 30
Participants
  At least one entry - fruit/veggie tracking: No | 7
  At least one entry - fruit/veggie tracking: Yes | 23
  At least one entry - Fitbit steps: No | 7
  At least one entry - Fitbit steps: Yes | 23

13. Primary Outcome: Intervention Feasibility Measures - Participant Engagement With Tracking
Description: Participant engagement with weekly diet/physical activity tracking measured by number of times participant engaged with the tracking feature at 6 months post-intervention
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who utilized tracking feature.
  Outcome for Arm 2 (Control/Delayed Intervention group) is not shown as this group did not have access to the FAITH! App and as such could not have participated in the described outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 30
Participants
  >=1 diet tracking entry | 23
  >=1 physical activity/steps tracking entry | 23

14. Primary Outcome: Number of Participants With and Without Engagement With Sharing Board
Description: Participant engagement with sharing board measured by number of posts per month by each participant at immediate post-intervention
Time Frame: Immediate post-intervention
Population: At least one app discussion board post. Number of participants analyzed reflects number of participants connected to app.
  Outcome for Arm 2 (Control/Delayed Intervention group) is not shown as this group did not have access to the FAITH! App and as such could not have participated in the described outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 30
Participants
  No | 26
  Yes | 4

15. Primary Outcome: Intervention Feasibility Measures - Participant Engagement With Sharing Board
Description: Participant engagement with sharing board measured by the number of participants sharing at least one discussion board post during the intervention
Time Frame: Immediate post-intervention
Population: App usage data as recorded by the device. Number of participants analyzed reflects number of participants connected to app.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 34 | 42
Participants | 5 | 10

16. Primary Outcome: Intervention Feasibility Measures - Participant Engagement With Modules
Description: App engagement as measured by the number of modules completed by the participants during the intervention. The number of participants who completed <5 and ≥5 modules (out of 10) was calculated.
Time Frame: Immediate post-intervention
Population: App usage data as recorded by the mobile device. Number of participants analyzed reflects number of participants connected to app.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 34 | 42
Participants
  <5 modules completed | 21 | 21
  ≥5 modules completed | 13 | 21

17. Primary Outcome: Intervention Feasibility Measures - App Usability
Description: App usability assesses four domains (Impact, Perceived usefulness, Perceived ease of use, User control) using the Health Information Technology Usability Evaluation Scale (Health-ITUES) instrument. 20 items are assessed, each on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). The overall Health-ITUES score was calculated as the mean of all 20 items, with each item being equally weighted. Possible total scores range from 1.0 (minimum) to 5.0 (maximum). A higher total sum indicates higher perceived usability of the technology measured at 6 months post-intervention.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 31 | 33
score on a scale
  Overall score | 4.2 (0.7) | 4.1 (0.6)
  Impact | 4.6 (0.6) | 4.2 (0.5)
  Perceived Usefulness: number analyzed (Participants) | 31 | 32
  Perceived Usefulness | 4.4 (0.7) | 4.1 (0.6)
  Perceived Ease Of Use | 3.9 (1.2) | 4.2 (0.8)
  User Control | 3.7 (1.0) | 3.9 (0.8)

18. Secondary Outcome: Smoking at Baseline as Assessed by Cigarette Smoking Status
Description: Self reported smoking status at baseline. Participants were asked to self-report current smoking status as "no" (non-smoker currently) or "yes" (current smoker). "Missing" category title indicates the survey response was unanswered.
Time Frame: Day 1
Population: Number of participants analyzed reflects number of participants who completed online questionnaire. Smoking status was not measured for change over time as it is a categorical variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 34 | 42
Participants
  No | 33 | 40
  Yes | 1 | 1
  Missing | 0 | 1

19. Secondary Outcome: Diet Self-Efficacy
Description: Changes from baseline to 6 months post-intervention in diet self-efficacy measured a 5-item scale to assess the participant's confidence in their ability to maintain a healthy diet when faced with common barriers. Each item is scored on a scale ranging from 0 (certain I cannot) to 100 (certain I can). A mean was calculated to obtain an overall score ranging from 0 (minimum) to 100 (maximum). The difference between the mean scores is calculated. A larger difference indicates larger change in self-efficacy for healthy eating. A negative change between baseline and 6 months post-intervention indicates worsened diet self-efficacy.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 29 | 28
score on a scale | 0.86 (21.19) | -5.30 (17.09)

20. Secondary Outcome: Diet Self-Regulation
Description: Changes from baseline to 6 months post-intervention in diet self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to eat healthier foods. Items are measured on a five-point scale from 1 (never) to 5 (always). A mean of all items is obtained and a difference between the scores is calculated. Higher change in scores indicate more change in use of self-regulation strategies to promote healthy eating.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 29 | 37
score on a scale
  Increase fruit/vegetable and grains | 0.43 (0.76) | 0.34 (0.70)
  Decrease fat and calories | 0.31 (0.69) | 0.18 (0.78)
  Plan and track nutrition | 0.68 (1.05) | 0.02 (1.03)

21. Secondary Outcome: Diet Social Support
Description: Changes from baseline to 6 months post-intervention in diet social support using the Social Support for Eating Habits Survey scale. This scale assesses the level of encouragement or discouragement from family and friends that participants received for adopting healthier eating habits. 5 questions were asked to assess the degree of encouragement and discouragement, separately, on a 5-point scale [from 1 (none) to 5 (very often)]. Each sub-item was summed to obtain a score ranging from 5 (lowest) to 25 (highest discouragement/encouragement). The change in level of diet social support was calculated from baseline to 6 months post-intervention. Higher scores indicate more change in social support for healthy eating.
Time Frame: 6 months post-intervention
Population: Number analyzed in specific rows may differ from overall number analyzed due to missing/unanswered responses from survey participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 30 | 28
score on a scale
  Family Encouragement | 1.33 (5.27) | 0.21 (4.21)
  Family Discouragement: number analyzed (Participants) | 29 | 27
  Family Discouragement | 0.28 (3.63) | 2.28 (5.10)
  Friend Encouragement: number analyzed (Participants) | 20 | 17
  Friend Encouragement | 0.50 (4.64) | 0.53 (4.21)
  Friend discouragement: number analyzed (Participants) | 20 | 17
  Friend discouragement | 0.61 (3.54) | 2.18 (5.82)

22. Secondary Outcome: Physical Activity Self-Efficacy
Description: Changes from baseline to 6 months post-intervention in physical activity self-efficacy measured using the Exercise Confidence Survey. The scale assesses the participant's confidence in their ability to exercise when faced with common barriers. 12 items are assessed, each on a 5-point scale ranging from 1 to 5. A mean of 8 items (Exercise confidence: Sticking to it) and 4 items (Exercise confidence: Making time for exercise) are obtained. The difference between baseline and 6 months post-intervention scores is calculated. A higher score indicates higher change in self-efficacy for physical activity.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 26 | 26
score on a scale
  Exercise confidence: Sticking to it | -0.12 (0.70) | -0.10 (0.64)
  Exercise confidence: Making time for exercise | -0.39 (0.85) | 0.00 (0.68)

23. Secondary Outcome: Physical Activity Self-Regulation
Description: Changes from baseline to 6 months post-intervention in physical activity self-regulation measured by the Health Beliefs Survey to assess strategies used in the past 3 months to increase their step count or physical activity levels. Items are measured on a 10-item five-point scale from 1 (never) to 5 (always). The mean of the ten items is obtained. The difference in the mean scores from baseline to 6 months post-intervention is calculated. Larger change in scores indicate more change in self-regulation.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 26 | 27
score on a scale | 0.56 (0.70) | 0.20 (0.74)

24. Secondary Outcome: Physical Activity Social Support
Description: Changes from baseline to 6 months post-intervention in diet social support using the Social Support for Exercise Survey scale. This scale assesses the level of encouragement or discouragement from family and friends that participants received for adopting healthier physical activity habits. 5 questions were asked to assess the degree of encouragement and discouragement, separately, on a 5-point scale [from 1 (none) to 5 (very often)]. Each sub-item was summed to obtain a score ranging from 5 (lowest) to 25 (highest discouragement/encouragement). The change in level of physical activity social support was calculated from baseline to 6 months post-intervention. Higher scores indicate more change in social support for physical activity. Family Participation was calculated as a sum of 10 items: 10 = low to 50 = high; Family Rewards/Punishment as a sum of 3 items: 3 = low to 15 = high; and Friend Participation sum of 10 items: 10 = low to 50 = high.
Time Frame: 6 months post-intervention
Population: Rows with numbers different than overall number analyzed are due to missing/unanswered survey responses from participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 26 | 36
score on a scale
  Family Participation | 3.12 (14.47) | -0.45 (7.97)
  Family rewards/punishment | 0.15 (2.17) | 0.28 (1.63)
  Friend Participation: number analyzed (Participants) | 21 | 30
  Friend Participation | 3.92 (9.22) | 1.61 (9.91)

25. Secondary Outcome: Psychosocial Measures - Religiosity/Spirituality
Description: Changes from baseline to 6 months post-intervention in Daily Spiritual Experiences Scale. Scores range from 1 to 6 (attendance), from 1 to 8 (prayer), and from 1 to 4 (religious coping), and from 6 to 36 (spirituality), with higher scores on each measure indicating greater religiosity.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 30 | 38
score on a scale | 0.07 (0.47) | 0.14 (0.46)

26. Secondary Outcome: Psychosocial Measures - Optimism
Description: Changes from baseline to 6 months post-intervention in life orientation test-revised scale. Scores range from 6 (least optimistic) to 24 (most optimistic). Participants respond to 3 positively worded items and 3 negatively worded items. Higher scores indicate more optimism.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 26 | 34
score on a scale | 0.23 (3.17) | -0.26 (3.18)

27. Secondary Outcome: Psychosocial Measures - Perceived Stress
Description: Changes from baseline to 6 months post-intervention in global perceived stress scale. The instrument measures global perceptions of stressful experiences over the prior 12 months in domains such as employment, legal issues, and racism/discrimination. Participants rate the severity of each domain according to a range from 1 (not stressful) to 3 (very stressful), with a total sum ranging from 0 to 24. Higher total scores indicate more perceived stress.
Time Frame: 6 months post-intervention
Population: Number of participants analyzed reflects number of participants who completed online questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Delayed Intervention/Control
Number analyzed (Participants) | 25 | 35
units on a scale | -0.08 (4.14) | -0.61 (5.76)

ADVERSE EVENTS:
Time Frame: Participants were monitored during 10 weeks of guided intervention, followed by a maintenance period of 6 months, for a total of approximately 9 months.
Arm/Group | Intervention | Delayed Intervention/Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 0/41 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03777709/Prot_SAP_000.pdf